CLINICAL TRIAL: NCT06706206
Title: The CACHE Study: Coronary Artery Care in HaEmophilia
Acronym: CACHE
Status: Recruiting | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Susie Shapiro, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 18218
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Haemophilia; Cardiovascular Diseases
MeSH Terms: conditions — Hemophilia A; Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Citrated blood samples for research markers of haemostasis/thrombosis, only retained for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational trial — Observational clinical trial. Participants will undergo cardiovascular risk assessment (clinical and blood tests) and coronary CT angiogram.
  These results will be compared to a control population without haemophilia (recruited as part of a different clinical trial).

SUMMARY:
The investigators will use state-of-the-art imaging to look at heart disease in people with haemophilia. Haemophilia is an inherited disorder in which blood does not clot properly because of lack of a key 'glue' blood component (chemicals known as factor VIII or IX). People with haemophilia are 40% less likely to die of heart disease, but it is not known exactly why this is. Understanding heart disease in people with haemophilia is important because better treatments for haemophilia mean that these patients are now living longer, but doctors still don't know if the risk for heart disease in these patients as they age is the same as that for the general population. If these processes are better understand (perhaps less blood clotting is actually protecting the heart from blockage-causing clots), scientists might be able to reduce the risk of heart attacks for everybody.

The UK's first photon-counting detector cardiac CT scanner generates detailed images of the heart and its blood vessels by counting individual X-ray photons. Together with artificial intelligence tools, it is possible to extract a lot of information from these images. As people age, fat is deposited in the vessels which supply blood to the heart which forms plaques. Plaques cause narrowing of the vessels, reducing blood flow to the heart, and can also burst (rupture), leading to a blood clot and heart attack. The new CT scan will show the type and amount of plaques, and quantify the risk of plaque rupture, in people with haemophilia; and the investigators will compare this to people without haemophilia.

Understanding the role of factor VIII/IX in heart attacks will improve management of heart disease in people with haemophilia, and may also lead to new prevention and treatment strategies that benefit heart health for everyone.

DETAILED DESCRIPTION:
Background and Rationale

Haemophilia, ageing and cardiovascular disease It is only relatively recently, due to the development of both effective and safe replacement therapies, that there is an aging population with haemophilia. This represents new challenges with respect to managing comorbidities. Cardiovascular disease (CVD) is the leading cause of death globally in the general population, and as people with haemophilia (PWH) age they are also at risk of developing CVD which poses particular challenges due to the opposing risks of bleeding, from haemophilia and antithrombotic treatments, versus thrombosis. Better understanding of the risks of atherosclerosis in PWH is crucial in order to best support aging PWH; and it has been identified as a research priority by patients and healthcare professionals.

Although mortality from cardiovascular disease in PWH has historically been about 40% less than the general population, it remains unclear whether this is because people with haemophilia develop atherosclerosis more slowly than the general population or whether deficiency of FVIII/FIX protects from formation of an occlusive thrombus at time of atherosclerotic plaque rupture. As FVIII is produced and stored within endothelial cells lining the blood vessels and FIX is produced in the liver, it may also be that FVIII and FIX deficiencies have different effects on the rates of atherosclerosis.

The most informative studies of atherosclerosis in PWH to-date used ultrasound to measure carotid and femoral intima-media thickness and computed tomography (CT) to derive coronary artery calcium scores. The first study measured carotid and femoral intima-media thickness (IMT) and brachial flow-mediated dilatation (FMD) as markers of atherosclerosis and endothelial dysfunction respectively in 51 obese PWH, and 42 obese and 50 matched non-obese male patients. All the PWH had haemophilia A (33% severe, moderate 16%, mild 50%), HIV was excluded, and the mean age was 50 +/-13 years. Carotid IMT was increased in obese as compared with non-obese subjects, but no difference was found in mean carotid and femoral IMT between obese PWH and obese control individuals. Thirty-five per cent of the obese PWH and 29% of the obese controls had an atherosclerotic plaque, irrespective of the severity of haemophilia. Brachial FMD was comparable between obese PWH and obese controls. The second study evaluated the presence and extent of atherosclerosis by coronary artery calcification score (CACS) derived from computed tomography and carotid IMT in 69 PWH (51 haemophilia A, 18 haemophilia B; 40% severe, 11% moderate, 49% mild). This again showed that CACS and carotid IMT were similar to controls and that the extent of atherosclerosis was related to traditional cardiovascular risk factors. Although these studies suggest PWH develop atherosclerosis at a similar rate to the general population; they are severely limited by the quality of the imaging techniques, patient numbers and relatively young patient age (average 50 years).

Cardiology guidelines recommend using a risk score to calculate cardiovascular risk over time and engaging patients in discussing modifiable risk factors. These scores have been used in PWH. A Dutch/UK cohort used both the QRISK(R)2 and SCORE algorithms. The predicted 10-year QRISK(R)2 risk was significantly higher in PWH than in the general population (8.9 vs. 6.7%), indicating more unfavourable cardiovascular risk profiles; and the increased risk became apparent after the age of 40 years. In contrast a study of 100 PWH in Europe compared to 200 aged-matched controls, found no significant difference in the 10-year cardiovascular mortality risk >10% between PWH and controls using SCORE. Other studies have looked at individual cardiac risk factors and PWH had higher rates of hypertension than expected for the general population. Critically whether the cardiac risk algorithm conveys the same actual CVD risk and is valid in PWH is not known.

Oxford University Hospitals has the ability to explore CVD risk and atherosclerosis in haemophilia with a proof of concept project due to having both a large haemophilia centre and the only UK photon-counting cardiac CT scanner.

Photon-counting cardiac CT

Coronary computed tomography angiography (CCTA) is a sensitive and widely used, non-invasive imaging modality for diagnosing coronary artery disease (CAD) and recent clinical guidelines have expanded its use as a first-line diagnostic tool in the management of chest pain of recent onset, suggestive of typical/atypical angina or non-anginal chest pain with electrocardiographic changes.

However, conventional CCTA identifies only anatomically significant coronary artery stenoses which are found in <50% of all patients referred for this test. Importantly, the majority of acute coronary syndromes are caused by unstable but non-obstructive atherosclerotic plaques, which cannot be identified by conventional CCTA or other non-invasive diagnostic tests detecting coronary luminal stenosis or stress-induced myocardial ischaemia. In the normal population, early detection of cardiovascular disease and subsequent optimisation has been associated with reduced cardiovascular mortality.

This has led to the development by our study investigators of the perivascular fat attenuation index (FAI or FAIPVAT), a novel imaging biomarker which detects vascular inflammation in the human coronary arteries using images from routine CCTA scans and is predictive of cardiovascular risk. The FAI relies on the discovery that inflammatory signals released by the diseased coronary artery, inhibit adipogenesis and trigger lipolysis in the perivascular adipose tissue (PVAT), shifting perivascular CT attenuation from the lipid towards that of the aqueous phase. Vascular inflammation is a driver of coronary atherosclerotic plaque formation, and a characteristic feature of atherosclerotic plaque rupture, leading to acute coronary syndromes including myocardial infarction. The causal role of inflammation in vascular disease pathogenesis has recently been documented by the CANTOS trial, which demonstrated that specific targeting of residual inflammatory risk improves clinical outcomes.

In the CRISP-CT study, recently published in the Lancet, our investigators demonstrated that FAIPVAT predicts all-cause and cardiac mortality over and above clinical risk factors and the current interpretation of CCTA. These findings are validated in two large and substantially different "real-life" prospective cohorts of patients undergoing clinically-indicated CCTA, one in Europe and the other in the United States, demonstrating similar predictive value.

Oxford University Hospitals has a newly-installed state of the art, photon-counting CT scanner, capable of performing CCTA to assess atherosclerotic burden and peri-vascular FAI. By incorporating an updated detector, single photons can be converted directly into electrical signals, removing the need for a two-step conversion process which is used in conventional CT scanners. This allows for higher resolution images than conventional CT at a given radiation exposure and therefore offers the opportunity to assess in detail the cardiovascular risk associated with haemophilia.

Oxford Haemophilia Centre

The Oxford Haemophilia Centre is one of the largest in the UK. The haemophilia team look after 190 PWH over the age of 40 years (range 40-88 years), of which 146 are over the age of 45 years, and 117 over the age of 50 years. Of PWH >45 years: 45 have severe haemophilia, 14 moderate haemophilia, 87 mild haemophilia; 77% have haemophilia A. Comorbidities are common and approximately 50% have hypertension and 7% atrial fibrillation. In those >65years, 6% have known ischaemic heart disease, 6% history of ischaemic stroke, and 4% peripheral vascular disease.

In order to help answer the question of whether PWH develop atherosclerosis at a similar rate to the general population with similar known cardiac risk factors, and whether there is a difference in the stability of the plaques, the investigators will use this state-of-the-art cardiac imaging technique to look in detail at atherosclerosis in aging patients with haemophilia and compare how this imaging data correlates with standard cardiovascular risk scores such as QRISK. As a comparison to general population, imaging data and standard cardiovascular risk factors will be compared to anonymised control scans from other studies at the University of Oxford with matching for age, gender, and exposure to cardiovascular risk factors (smoking, hypertension, high cholesterol, diabetes, family history). These data could pave the way for future multi-centre clinical studies with increased numbers of PWH (especially through close regional haemophilia centres and potentially reducing age of screening), extension to other common bleeding disorders such as von Willebrand disease, and ultimately impact on clinical care for people with bleeding disorders (cardiac screening); as well as further translational research studies into the role of factor VIII and factor IX in the pathogenesis of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to give informed consent for participation in the study.
* Male, aged 45 years or above (no upper age limit).
* Haemophilia A or B with Factor VIII/IX less than 40% (0.40 IU/ml).

Exclusion Criteria:

* Participants unable or unwilling to give informed consent.
* Participants unable to understand the English language.
* Participants unable or unwilling to attend for the necessary scans and investigations.
* Patients with absolute contra-indications to CT imaging will be excluded from the study. This includes:

  * Any known contraindications to CT iodinated Contrast.
  * Significant renal impairment (eGFR <30 ml/min).
* Any other medical conditions which would influence the reliability of the study results determined by the investigators.

Ages: 45 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have a diagnosis of haemophilia A or B. Participants must be 45 years or older.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of coronary artery disease detected by coronary CT angiogram among people with haemophilia (PWH) versus control group. | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  This is the primary outcome within the primary objective 'to determine whether coronary artery disease (presence of atherosclerotic plaques, type, burden, fat attenuation index (FAI)) in PWH is similar to the control population matched for standard cardiac risk factors.'

SECONDARY OUTCOMES:
Quantitative analysis of the volume of each plaque component (calcified, non-calcified, low-density plaques) among people with haemophilia (PWH) compared to control group. | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  This is the secondary outcome within the primary objective 'To determine whether coronary artery disease (presence of atherosclerotic plaques, type, burden, FAI) in PWH is similar to the control population matched for standard cardiac risk factors.'
Quantitative analysis of fat attenuation index (FAI) among PWH compared to control group. | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  This is the secondary outcome within the primary objective 'To determine whether coronary artery disease (presence of atherosclerotic plaques, type, burden, FAI) in PWH is similar to the control population matched for standard cardiac risk factors.'

OTHER OUTCOMES:
Secondary Objectives (1a): Subgroup analysis to evaluate the influence of haemophilia severity and type on the occurrence of coronary artery disease as detected by CCTA. | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  Occurrence of coronary artery disease detected by CCTA among PWH vs control group.
Secondary Objectives (1b): Subgroup analysis to evaluate the influence of haemophilia severity and type on the volume of each plaque component. | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  Quantitative analysis of the volume of each plaque component (calcified, non-calcified, low-density plaques)
Secondary Objectives (1c): Subgroup analysis to evaluate the influence of haemophilia severity and type on the fat attenuation index (FAI). | Participant demographics and cardiovascular risk factors to be collected at enrolment for matching PWH and control group. Photon counting CCTA to be performed at enrolment for prevalence of CAD, and quantitative analyses in the secondary outcome.
  Quantitative analysis of fat attenuation index (FAI) Score for quantification of coronary inflammation.
Secondary Objectives (2) : To understand the underlying pathophysiological mechanisms and impact of haemophilia and atherosclerosis. | Blood tests at enrolment for research analysis of inflammatory and prothrombotic biomarkers.
  Inflammatory and prothrombotic blood biomarkers; comparison with CCTA results.
Secondary objectives (3): To assess actual cardiovascular events at 5 years, and model how this compares to general population risk prediction models. | Review of clinical cardiovascular history 5 years after enrolment.
  Cardiac death and other major adverse cardiac events (ischaemic cardiac events (angina, acute coronary syndromes), new onset heart failure, stroke) will be collected for the haemophilia population and will be compared to the predicted 5 year event rate based on baseline QRISK/CCTA and the actual 5 year event rate of the control population.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Haemophilia and Thrombosis Centre, Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided